CLINICAL TRIAL: NCT06873282
Title: Randomized, Double-blind, Placebo-controlled Phase 2 Trial of ТВ/Flu-05Е Intranasal Vector Vaccine for the Prevention of Tuberculosis Infection in BCG-vaccinated Volunteers Aged 18-50 Years
Brief Title: Phase 2 Study of the ТВ/Flu-05Е Tuberculosis Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Research Institute of Influenza, Russia (Other)
Collaborators: Pavlov First Saint Petersburg State Medical University (Other); St. Petersburg City Polyclinic No. 34 (Unknown)
Responsible Party: Principal Investigator, Tatyana Zubkova, Head of the clinical department, Research Institute of Influenza, Russia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ВПТ-2-06/2023
Record Dates: First submitted 2025-03-06; First posted 2025-03-12 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2023-11

CONDITIONS: Tuberculosis
Keywords: Tuberculosis vaccine; BCG boost; influenza vector; mucosal vaccine
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TB/Flu-05E (Experimental): Single dose of TB/Flu-05E vector vaccine
  Interventions: Biological: TB/Flu-05E
- Placebo (Placebo Comparator): Single dose of Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: TB/Flu-05E — Participants will receive single intranasal injection of TB/Flu-05E vaccine in 0.5 ml, containing 7.7 lg EID50 of A/H1N1pdm09 recombinant attenuated influenza vector with modified NS gene, encoding for the TB10.4 and HspX antigens of M. tuberculosis
  Arms: TB/Flu-05E
Other: Placebo — Participants will receive single intranasal injection of physiological buffer in 0.5 ml
  Arms: Placebo

SUMMARY:
The aim of the study is to investigate immunogenicity and safety of the TB/Flu-05E single-dose intranasal vaccine for the prevention of Tuberculosis infection in BCG-vaccinated Volunteers aged 18-50 years

DETAILED DESCRIPTION:
Study includes 160 participants aged 18 to 50, randomized at 3:1 ratio, to receive single intranasal dose of TB/Flu-05E vaccine or placebo, correspondingly. Duration of the study for each participant is about 4 months (no more than 114 days).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy BCG-vaccinated men and women aged 18 to 50 years
2. Availability of signed informed consent
3. Diagnosed "healthy" according to the data of standard clinical, laboratory and instrumental examination methods, with the absence of clinically significant changes. Participants with chronic conditions that do not require special treatment, such as diabetes mellitus, hypertension, or heart disease, are eligible to participate in this study if the investigator considers the participant's condition to be medically stable
4. The ability and willingness to make entries in the diary of self-observation, as well as to carry out all the visits foreseen in the study for control medical observation
5. Consent of study participants to use effective contraceptive methods throughout their participation in the study. In this study, volunteers can use the following methods of contraception:

   * Barrier methods:

     * male condom and spermicide
     * cervical cap and spermicide
     * vaginal diaphragm and spermicide
   * Intrauterine device
   * Hormonal intrauterine device
   * Hormonal contraceptives:

     * hormonal implants
     * hormone injections
     * combined oral contraceptives
     * mini-pill
     * contraceptive patch
   * Abstinence from sexual activity.
6. Body weight ≥ 50 kg
7. Negative test for alcohol in exhaled air
8. Values of the complete blood count and biochemical blood analysis (during the screening) within 0.9*reference range lower limit and 1,1 * reference range upper limit
9. Negative tests for HIV, hepatitis B, hepatitis C, and syphilis
10. Absence of pathological changes on the chest X-ray (fluorogram of the lungs).

Exclusion Criteria:

1. Participation in another clinical study within three months prior to the start of the current study; planning to participate in another study during the current study period
2. Clinical, radiological or laboratory signs of active or previously transferred tuberculosis of any localization.
3. Existence in the past or present of contact with patients with any form of tuberculosis (at home, at work, in the circle of friends and acquaintances)
4. Tuberculous infection confirmed by the TB-FERON IGRA laboratory test
5. Immunization with BCG within six months prior to enrollment in the current study
6. Contact with COVID-19 patients within 14 days prior to the start of the clinical study
7. Positive rapid test result for SARS-CoV-2 antigen
8. Immunization with any other non-study vaccine product within three weeks prior to enrollment in the current study, or refusal to postpone such until the end of the three-week period after completion of the current study
9. Regular use of nasal irrigation therapy during the last six months prior to enrollment in the current study or episodic use of the above method of treatment in the two weeks prior to the screening
10. History of frequent nosebleeds (>5) during the year prior to the current study
11. Features of the nasal anatomy that may complicate intranasal administration of the study drug.
12. Surgical interventions or traumatic injuries in the sinus area, paranasal sinuses, or traumatic injuries of the nose within a month before screening
13. Symptoms of acute respiratory disease, including fever, or other acute illness at the time of screening or within two weeks prior to screening
14. Treatment with immunoglobulins or other blood derived medications in the three months prior to screening or planning such treatment during the period of participation in the current study
15. History of bronchial asthma
16. Hypersensitivity and the presence of severe allergic reactions, including Quincke's edema, anaphylactic shock after the previous administration of any vaccine
17. History of wheezing after previous immunization with live influenza vaccine
18. Other adverse events after immunization (fever above 40°C, syncope, non-febrile convulsions, anaphylaxis) when there is a minimal likelihood that they are associated with a previous administration of any vaccine
19. Suspicion of hypersensitivity to any component of the study vaccine, including egg protein
20. Acute or chronic clinically significant lung, cardiovascular, hepatic, endocrine, neurological, or psychiatric disorders, or impaired renal function identified by history, physical examination, or clinical laboratory findings that, in the opinion of the investigator, may influence the outcome of the study
21. History of oncological diseases
22. History of thrombocytopenic purpura or bleeding disorders
23. History of convulsions
24. Chronic alcohol dependence or chronic use of illicit drugs, drug abuse
25. Claustrophobia and social phobia according to history and / or available medical records
26. Inability to read Russian; inability or unwillingness to understand the essence of the study
27. Military personnel undergoing military service on conscription
28. Special diet (eg, vegetarian, vegan, salt-restricted) or lifestyle (night work, extreme physical activity)
29. Any condition that, in the opinion of the investigator, may increase the risk to the health of a volunteer participating in the study or affect the results of the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2023-12-13 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-04-11 (Actual)

PRIMARY OUTCOMES:
Level of TB antigen-specific cytokine producing T-cells | Days 1, 7, 21
  Change from baseline in the level of cytokine producing T-cells upon in vitro stimulation of PBMC with M. tuberculosis peptide epitopes (TB10.4, HspX) measured by FACS/ELISPOT
Level of TB antigen-specific cytokine release in whole blood assay | Days 1, 7, 21
  Change from the baseline of the cytokine concentration in whole-blood cytokine release assay upon in vitro stimulation with M. tuberculosis peptide epitopes (TB10.4, HspX) measured in ELISA

SECONDARY OUTCOMES:
Number of participants with local and systemic adverse events (AEs) and serious adverse events (SAEs) | Throughout the study, average 4 months
  Adverse events (AEs) and serious AEs (SAEs), both vaccine related, and non-vaccine related. AEs/SAEs of particular importance: - Immediate AEs (allergic reactions) occurring within two hours of vaccination;
  - Post-vaccination reactions (anticipated clinical manifestations of a local and systemic nature), usually due to intranasal vaccination between two hours and the next 7 days after vaccination
Percent of participants with T-cell response to M. tuberculosis antigens | Days 7, 21
  Relative number of participants with T-cell response to the M. tuberculosis antigens (TB10.4 or HspX) in any of the tests (FACS/ELISPOT, whole blood cytokine release assay) at any of the study days
Level of TB antigen-specific IgG antibody in serum | Days 1, 21, 111±3
  Change from the baseline in the level of TB10.4 and HspX specific IgG antibody measured in ELISA in serum
Level of B-cell and Tfh-cell populations | Days 1, 7, 21
  Change from the baseline in the relative amount of B-cell and Tfh-cell populations measured by FACS
Level of mucosal IgA antibody in nasal secret | Days 1, 21
  Change from the baseline in the level of IgA antibody measured in ELISA in nasal secret
Level of influenza-specific cytokine producing T-cells | Days 1, 7, 21
  Change from baseline in the level of cytokine producing T-cells upon in vitro stimulation of PBMC with influenza antigen measured by ICS/ELISPOT
Influenza specific systemic antibody immune response | Days 1, 21, 111±3
  Change from baseline in the titer of influenza specific antibodies in serum measured in hemagglutination inhibition/microneutralization assay

CONTACTS AND LOCATIONS:
Overall Officials: Marina Stukova, Dr, Study Director — Smorodintsev Research Institute of Influenza
Locations (3):
- Russia (3):
  - Pavlov First Saint Petersburg State Medical University, Saint Petersburg
  - Smorodintsev Research Institute of Influenza, Saint Petersburg
  - St. Petersburg City Polyclinic No. 34, Saint Petersburg

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication will be available
Access Criteria: IPD will be available upon reasonable request to Study Director. Once the request is approved, the data can be transferred via a secure online platform